CLINICAL TRIAL: NCT00538265
Title: Evaluation of the Benefit of Antithymocyte Induction Therapy on Hepatic Fibrosis in de Novo Hepatitis C Virus Liver Transplant Patients.
Brief Title: Benefit of Immunoprophylaxis on Fibrosis to Reduce Viral Load After Liver Transplantation
Acronym: BEFIRTH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: LLAU ME, University Hospital Toulouse
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0404003
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Liver Transplantation
Keywords: liver transplantation, hepatitis C virus, immunoprophylaxis
MeSH Terms: conditions — Hepatitis C | interventions — Tacrolimus; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): tacrolimus + steroids
  Interventions: Drug: tacrolimus
- B (Experimental): ATG+ tacrolimus without steroids in maintenance therapy
  Interventions: Drug: tacrolimus, ATG
- C (Experimental): ATG+ Mycophenolate Mofetil + tacrolimus a reduced dosage without steroids in maintenance therapy
  Interventions: Drug: ATG+mycophénolate mofétil+tacrolimus

INTERVENTIONS:
Drug: tacrolimus — Tacrolimus started at 0.50 mg/kg b.i.d. starting at D0, by nasogastric tube and then 1 to 2 hours before meals. The dose of tacrolimus will be adjusted as soon as possible to obtain trough concentrations of the product between 10 and 20 µg/L between D0 and 6 months and then between 8 and 15 µg/L after 6 months
  Other Names: PROGRAF
  Arms: A
Drug: tacrolimus, ATG — immunoprophylaxis allowing sparing of steroids in maintenance therapy combining induction therapy with 3 injections of antithymocyte globulins (ATG) (1.5 mg/kg/d at D0, D2 and D4) and tacrolimus at usual dosage.
  In this group of patients, the first injection of ATG will be infused over a period of at least 6 hours and will be started as soon as vascular anastomosis has been completed. It will be preceded by an injection of 3 mg/kg/d methylprednisolone. The second injection of ATG at D2, post transplantation will also be infused over 6 hours and will be preceded by an injection of 1 mg/kg methylprednisolone, and then subsequently steroids will be excluded from the treatment. The third and last injection at D4 post transplantation will be administered over a 6-hour period but will not be preceded by steroids.
  In this study arm, tacrolimus will be administered as in arm (A)
  Other Names: Thymoglobuline
  Arms: B
Drug: ATG+mycophénolate mofétil+tacrolimus — immunoprophylaxis allowing sparing of steroids in maintenance therapy combined with mycophenolate mofetil, at an initial dosage of 2 grams a day, and then adjusted to safety and tolerability in such a way so as to maintain PMN ≥ 750/mm3, and platelet counts ≥ 30000/mm3.
  In this study arm, the patients will receive the same doses of ATG and steroids (and according to the same methods) as in arm B. Tacrolimus started at 0.05 mg/kg b.i.d. starting at D0 by nasogastric tube and then 1 to 2 hours before meals. In this study arm, the tacrolimus dose will be reduced: targeted trough concentrations will be between 7 and 12 µg/L between D0 and 6 months and then between 3 et 7 µg/L after 6 months.
  Other Names: Mycophénolate mofétil = Cellcept
  Arms: C

SUMMARY:
An open-label randomized multicenter clinical study comparing three regimes of immunosuppression : (A) tacrolimus and steroids, (B) antithymocyte induction therapy and full dose of tacrolimus, (C) antithymocyte induction therapy with mycophenolate mofetil and a reduced dose of tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* patients who received a first liver transplantation,
* presenting with a qualitative or quantitative PCR positive for hepatitis C virus at time of transplantation, whatever the transaminase activity,
* Women of childbearing potential with a negative pregnancy test,
* Male or female patients who agree to use an effective method of contraception,
* patients who signed a written informed consent form to participate in the study,
* patients who are compliant and likely to follow the visits specified by the study protocol

Exclusion Criteria:

* • Preoperative serious renal impairment (serum creatinine levels > 200 µmol/l),

  * repeat transplantation,
  * multiple organ transplantation,
  * transplantation performed with an organ transplant obtained from a living donor or a reduced or shared organ grafts,
  * serious concomitant disorder,
  * positive serology for HBs antigen or HIV positive at time of enrollment,
  * previous history of nonhepatic cancer (except for localized skin cancer),
  * presence of a hepatocellular carcinoma, for which the primary lesion exceeds 5 cm or is complicated by portal thrombosis or metastatic disease,
  * an investigational product or therapy administered less than one month before entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-05; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be degree of fibrosis = Ishak's histological score of hepatic biopsy at 1 year | 1 year

SECONDARY OUTCOMES:
• Ishak's degree of activity | 1 year
Ishak's degree of fibrosis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rostaing Lionel, PhD, Principal Investigator — University Hospital, Toulouse; Calmus Yvon, PhD, Principal Investigator — UHCochin, Paris
Locations (8):
- France (8):
  - Hopital Pellegrin Tripode, Bordeaux
  - La CONCEPTION hospital, Marseille
  - Hopital Saint-Eloi, Montpellier
  - Hopital de L'Archet, Nice
  - Hôpital Cochin, Paris
  - Hôpital Pontchaillou, Rennes
  - University Hospital, Toulouse
  - Hopital Paul Brousse, Villejuif